CLINICAL TRIAL: NCT00086632
Title: An Open-Label, Phase II Study of Ovarex® MAb-B43.13 as an Adjuvant Treatment to Platinum-Based Front-Line Chemotherapy of Advanced Epithelial Carcinoma of Ovarian, Tubal, or Peritoneal Origin
Brief Title: Study of Ovarex® (Oregovomab) MAb With Front-Line Chemotherapy for Ovarian Cancer Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed by sponser
Sponsor: Unither Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVA-Gy-18
Record Dates: First submitted 2004-07-07; First posted 2004-07-09 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2006-01

CONDITIONS: Ovarian Cancer
Keywords: oregovomab; ovarex; ovarian cancer; ovary; ovarian carcinoma; front-line
MeSH Terms: conditions — Ovarian Neoplasms | interventions — oregovomab

INTERVENTIONS:
Drug: oregovomab

SUMMARY:
An experimental treatment with OvaRex® MAb-B43.13 (oregovomab), called immunotherapy is being tested in ovarian cancer patients. Immunotherapy causes the body's defenses to react against cancer cells. The purpose of this research study is to determine if immunotherapy with oregovomab can create an immune response and enable the body to fight the disease and help ovarian cancer patients live longer. Patients with a possible diagnosis of ovarian cancer will be screened for study participation pre-surgery and, if eligible, will receive oregovomab during front-line chemotherapy treatment for ovarian cancer and quarterly for about a year following chemotherapy. Patients who experience disease progression will be discontinued from oregovomab therapy. Patients will also have urine, blood and tissue samples collected to assess the immune response to oregovomab.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of primary peritoneal carcinoma or epithelial ovarian carcinoma, Stage III - IV, expressing the tumor-associated antigen CA125 as measured by a serum CA125 level ≥ 35 U/mL and tumor tissue which has been demonstrated by immunohistochemical methods to express CA125. All patients must provide primary tumor (and lymph node and ascites samples, if available) samples for cellular immunology assays and characterization
* A functional performance status of ≤2 on the ECOG scale
* Are randomized into the study no more than eight (8) weeks postoperatively
* Have an expected survival of at least 6 months
* Age less than or equal to 80 years of age
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care

Exclusion Criteria:

* Have received radiotherapy or chemotherapy
* Have circumstances at the time of entry onto the protocol would not permit completion of study or require follow-up
* Have other invasive malignancies, with the exception of non-melanoma skin cancer and carcinoma in situ of the cervix, who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Have significant cardiovascular abnormalities [uncontrolled hypertension, Congestive Heart Failure (CHF) New York Heart Association (NYHA) Classes II-IV, see Appendix C), uncontrolled angina, myocardial infarction within the past six months or uncontrolled arrhythmias]. Patients with evidence of abnormal cardiac conduction (e.g. bundle branch block, heart block) are eligible if their disease has been stable for the past six months
* Have an active autoimmune disease (e.g., rheumatoid arthritis, Systemic Lupus Erythematosus (SLE), ulcerative colitis, Crohn's Disease, MS, ankylosing spondylitis) requiring active immunosuppressive therapy
* Have a known allergy to murine proteins or have had a documented anaphylactic reaction to any drug
* Are being chronically treated with immunosuppressive drugs such as cyclosporin, Adrenocorticotrophic Hormone (ACTH), or systemic corticosteroids
* Have a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; patients who have acquired, hereditary, congenital immunodeficiencies, Human Immunodeficiency Virus, or status post splenectomy
* Have an uncontrolled disease (e.g. deteriorating renal function or nephropathy, active hepatitis, etc.) other than cancer. Patients with chronic diseases that are well controlled (e.g., diabetes mellitus, hypertension) are eligible
* Are taking mono-amine oxidase inhibitors or who have other contraindications to the use of pressor agents (e.g. epinephrine)
* Are unable to read or understand, and/or unwilling to sign a written consent form which must be obtained prior to surgery and prior to treatment Surgery
* Patients will not be required to undergo second-look surgery (such surgery will be at the option of the investigator)
* If patients undergo a second surgical procedure for a clinically indicated circumstance, an interval tumor sample with ascites and lymph node (if available) should be obtained, if present, for immunological evaluation and provided to the study tissue bank

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-07; Study Completion 2007-12 (Actual)